CLINICAL TRIAL: NCT07389473
Title: An Observational Study to Evaluate the Effects of Long-term Use of Psychotropic Medications on Eye Movement Patterns With the Gaize Device
Brief Title: Evaluate the Effects of Long-term Use of Psychotropic Medications on Eye Movement Patterns With the Gaize Device
Acronym: Rx Meds Gaize
Status: Recruiting | Type: Observational
Sponsor: Gaize (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-GPHPV-01
Record Dates: First submitted 2025-08-20; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: ADHD; Depression Disorders; Mood Disorders; Anxiety Disorder Generalized; Bipolar Disorder (BPD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Mood Disorders; Generalized Anxiety Disorder; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Participants will be recruited through local participants. Local psychiatrists will be enlisted to inform eligible patients about the research. Psychiatrists will disseminate information via study flyers displayed in their offices and through direct conversation with patients during appointments. This approach ensures informed and voluntary participation from individuals familiar with the psychiatric medication regimen, aligning with ethical research practices and privacy regulations. Potential participants' eligibility will be assessed based on predefined inclusion and exclusion criteria. If individuals meet these criteria and express interest, they will be provided with information about the study's objectives, potential risks, and benefits.
  Interventions: Drug: Prescription Psychotropic Medications
- Control Group: We will recruit control group participants by posting up flyers to the general population through community bulletin boards, social media, and local community health centers. These participants will be matched to our patient group by age, sex, and other relevant demographic factors but will not be taking psychotropic medications. Interested individuals will undergo a screening process to ensure they meet the specific criteria for the control group. To maintain transparency and informed consent, all participants, both in the study and control groups, will receive consent forms. Those willing to participate will have the opportunity to review and sign these forms.
  Interventions: Drug: Prescription Psychotropic Medications

INTERVENTIONS:
Drug: Prescription Psychotropic Medications — Currently using a psychiatric medication as prescribed by a healthcare professional for longer than 3 months.

SUMMARY:
The study aims to verify if the Gaize ocular device can effectively identify eye movements indicative of prescribed psychotropic medication usage by employing Drug Recognition Expert (DRE) testing protocols within a controlled virtual environment.

DETAILED DESCRIPTION:
The use of psychotropic (psychiatric) medications for various psychiatric disorders is a common practice. Long-term use of such medications necessitates monitoring due to potential side effects, including ophthalmic issues (1). The Gaize VR headset represents a novel approach to monitoring these effects by utilizing Drug Recognition Expert (DRE) testing methods to detect eye movements associated with substance use.

Psychotropic medications have been associated with a range of visual and oculomotor side effects, which can impact patient safety and quality of life (2). The prevalence of these effects in long-term users is not fully characterized in the literature, and traditional methods of assessment may miss subclinical alterations in eye movement or function. Eye movement patterns are altered predictably by the use of various substances, such as cannabis, alcohol, and other psychoactive drugs. DRE protocols utilize oculomotor tests to infer recent drug use (3). These protocols are, however, often subjective and require trained personnel to administer, leading to potential variability in assessment and risk of false positives. Advances in virtual reality technology have allowed for more precise and controlled assessment of eye movements. VR headsets can isolate and measure specific eye movement parameters, potentially providing a more accurate and objective measure of oculomotor function and impairment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65, having given written informed consent to participate in the research trial.
* Currently using a psychiatric medication as prescribed by a healthcare professional for longer than 3 months.
* Normal or corrected to normal vision using either glasses or contact lenses, or surgery.

Exclusion Criteria:

* Enrolled in, or participated in another clinical trial within 30 days before the study
* Having a prosthetic eye, missing eye, or wearer of an eye patch LASIK or other eye surgery within the prior 21 days.
* Had your eyes dilated by a medical doctor in the previous 24 hours.
* Photosensitive epilepsy
* Diagnosed with clinical blindness
* Medical Conditions: Participants with medical conditions or medications that could significantly affect cognitive and motor functions are excluded. Participants with conditions such as Glaucoma, macular degeneration, cataracts, lazy eye (amblyopia), or optic neuritis, or genetic anisocoria (unequal pupil size) will be excluded.
* Current or past head inject/ traumatic brain injury (TBI)
* Pregnancy: Pregnant individuals will be excluded from the study due to the potential risks associated with psychiatric medications.
* History of Severe Motion Sickness: Participants with a history of severe motion sickness in VR environments may be excluded, as they may not tolerate the VR headset well.
* Potential participants who are unable to provide consent for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant population is limited to the city of Philadelphia, PA
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Collection of Ophthalmic Data | 1 Day
  Accuracy of the Gaize device in detecting eye-movement metrics consistent with prescribed psychotropic medication use, as determined by Drug Recognition Expert (DRE) testing protocols in a controlled virtual environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaize, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hartman RL, Richman JE, Hayes CE, Huestis MA. Drug Recognition Expert (DRE) examination characteristics of cannabis impairment. Accid Anal Prev. 2016 Jul;92:219-29. doi: 10.1016/j.aap.2016.04.012. Epub 2016 Apr 22. PMID 27107471
- [Background] Williams R, Hui A. Common systemic medications that every optometrist should know. Clin Exp Optom. 2022 Mar;105(2):149-156. doi: 10.1080/08164622.2021.1945409. Epub 2021 Aug 18. PMID 34407728
- [Background] Mahal P, Suthar N, Nebhinani N. Spotlight on Oculogyric Crisis: A Review. Indian J Psychol Med. 2021 Jan;43(1):5-9. doi: 10.1177/0253717620942096. Epub 2020 Sep 3. PMID 34349300